CLINICAL TRIAL: NCT05872282
Title: Feasible Study on a New Technique of ZIPPER Aortic Arch Stentgraft System in the Treatment of Aortic Arch Disease
Brief Title: Percutaneous Endovascular Arch Repair Trial (PEART) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Collaborators: Wayne W.Zhang , Seattle，Washington，USA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZIPPER V1.0
Record Dates: First submitted 2023-05-09; First posted 2023-05-24 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-05

CONDITIONS: Aortic Diseases
Keywords: Aortic Arch; Dissection; aneurysm
MeSH Terms: conditions — Aortic Diseases; Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZIPPER aortic arch stentgraft system (Experimental)
  Interventions: Device: ZIPPER aortic arch stentgraft system

INTERVENTIONS:
Device: ZIPPER aortic arch stentgraft system — The ZIPPER aortic arch stentgraft system consists of the arch mainbody stentgraft system, the branch artery stentgraft system and the thoracic extension stentgraft system.

SUMMARY:
This study is the feasible study on a new technique of ZIPPER aortic arch stentgraft system

DETAILED DESCRIPTION:
The feasible study of ZIPPER aortic arch stentgraft system is a prospective, multicenter, single arm trial, which will enroll a total of 24 patients. The goal of this study is to evaluate the safety and efficacy of ZIPPER aortic arch stentgraft system in the treatment of patients with aortic arch disease, included aortic arch dissections, aneurysms, residual dissection following ascending aorta surgical operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years old
2. Patients diagnosed with aortic arch disease requiring intervention, including non-A-non-B aortic dissection, or residual dissection after type A ascending aortic repair; aortic arch aneurysms.
3. Patients with suitable vascular conditions, including:

   1. Ascending aorta (including surgical graft) length greater than 30 mm (from the aortic sinusoid junction to the proximal cardiac margin of the innominate artery).
   2. Proximal anchoring zone diameter ≥ 24 mm and ≤ 47 mm;
   3. Proximal anchoring zone length ≥ 20 mm;
   4. Innominate artery, left common carotid artery and left subclavian artery diameter ≤ 24 mm and ≥ 7 mm, length ≥ 20 mm；
   5. Suitable arterial access for endovascular interventional treatment;
4. Patients able to understand the purpose of the trial, participate in the trial voluntarily with informed consent form signed by the subject him/herself or his or her legal representative, and willing to complete follow-up visits as required under the protocol.
5. Evaluated by at least two investigators that the subjects are high-risk patients with more complications, poor general condition, high risk of deep hypothermic circulatory arrest, and not suitable for total arch replacement and other surgical procedures.

Exclusion Criteria:

1. Previously received open surgery or endovascular intervention for descending aorta or abdominal aorta;
2. Infectious aortic disease, takayasu arteritis, Marfan syndrome (or other connective tissue diseases );
3. Patients that have experienced systemic infection within past three months;
4. Neck surgery was performed within past three months;
5. Patients with severe stenosis, calcification, thrombosis or tortuosity in the brachiocephalic trunk, left common carotid artery or left subclavian artery;
6. Patients with intestinal necrosis and lower limb ischemic necrosis;
7. Paraplegic patients;
8. Heart transplant patients;
9. Patients that have suffered MI or stroke within past three months;
10. Patients with Class IV heart function (NYHA classification) or LVEF<30%
11. Active peptic ulcers or upper gastrointestinal bleeding occurring within the past three months;
12. Hematological abnormality, defined as follows: Leukopenia (WBC < 3 × 109/L), anemia (Hb < 90 g/L); coagulation dysfunction, thrombocytopenia (PLT count< 50 × 109/L);
13. Patients with renal insufficiency， serum creatinine > 150 umol/L (or 3.0 mg/dl) and / or end-stage renal disease requiring dialysis, shall be determined by the investigator after a comprehensive analysis;
14. Patients with severe liver dysfunction: ALT or AST exceeding 3 times the upper limit of norma, serum total bilirubin (STB) exceeds 2 times the upper limit of normal;
15. Patients who are allergic to contrast agents;
16. Patients that are pregnant or breastfeeding;
17. Patients with severe comorbidities who cannot tolerate anesthesia and surgery;
18. Patients with a life expectancy of less than 12 months;
19. Patients currently participating in other drug or device study;
20. The investigator assessed that the patient was ineligible for the study for other diseases or abnormalities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
Freedom from major device/procedure-related adverse events within 30 days post-operation. | 30 days after intervention
  Device or procedure related major adverse events included: stroke, respiratory failure, pericardial tamponade, dissection or aneurysm rupture, paraplegia, stent occlusion, fracture, migration, access vessel thrombosis or rupture, conversion to open surgery, death.

SECONDARY OUTCOMES:
Immediate postoperative technical success. | immediately after intervention
  Immediate technical success is defined as successful delivery of the aortic and branching stent graft conveyors to their predetermined positions, accurate positioning and successful deployment of the stent, safe removal of the delivery device outside the body, absence of Type I and III endoleaks on angiography at the end of the procedure , and patent branch stents.
Incidence of Type I or Type III endoleaks. | 1 month, 6 months and 12 months post-intervention
  Endoleak evaluated by DSA or CTA during operation and at 1 month, 6 months and 12 months after operation. Intraoperative endoleaks that were treated with adjuvant therapy were not documented. Endoleaks occurring in the same subject after completion of the procedure, and that were not treated at different visits, are counted as once.
Incidence of aortic arch stent graft migration. | 1 month, 6 months and 12 months post-intervention
  CTA will be performed at 1, 6, and 12 months after operation to determine if the stent has migrated, and evaluations will be recorded for both the main and branch stents. Migration is defined as the main and branched stents migrate more than 10 mm at postoperative follow-up compared with that 1 month post-intervention.
Postoperative branch vessel patency rate. | 1 month, 6 months and 12 months post-intervention
  CTA examinations will be performed at 1, 6, and 12 months post-operation to evaluate branch vessel revascularization and whether there is occlusion, stenosis, or stent thrombosis.
Results of aortic remodeling after aortic dissection surgery | 1 month, 6 months and 12 months post-intervention
  CTA examinations will be performed at 1, 6, and 12 months post-operation to evaluate results of aortic remodeling, including the expansion of the true lumen and the thrombosis of the false lumen at the coverage of the aortic dissection vascular stent to determine whether the blood vessel is successfully remodeled.
Progression control of aortic aneurysm | 1 month, 6 months and 12 months post-intervention
  CTA examinations will be performed at 1, 6, and 12 months post-operation to evaluate results of progression control of aortic aneurysm. The maximum diameter of aortic aneurysm increases by ≤ 5 mm after 12 months of CTA examination compared with that before surgery.
Incidence of surgically induced de novo aortic dissection converted to open-heart surgery or secondary intervention. | within 12 months post-intervention
  Whether or not the patient experienced surgically induced de novo aortic dissection converted to open-heart surgery or secondary intervention will be determined.
Aortic-related mortality at 12 months post operation. | within 12 months post-intervention
  Refers to death caused by aortic rupture or endovascular treatment.
All-cause mortality and major stroke within 12 months post-procedure. | within 12 months post-intervention
  All-cause mortality includes cardiac death, non-cardiac death, and unexpected death. Major stroke is defined as a modified Rankin score (mRS) ≥ 2 at 90 days after stroke onset.
Incidence of severe adverse events. | within 12 months post-intervention
  Refers to an event that occurs during the clinical trial that results in mortality or serious deterioration in patient health, including a fatal illness or injury, a permanent defect in body structure or body function, or an event that requires medical or surgical intervention to avoid one or more permanent defects in body structure or body function.
Incidence of device-related adverse events. | within 12 months post-intervention
  Device-related adverse event refers to an adverse medical event related to the use of test device during the clinical trial. However, a distinction should be made with respect to normal postoperative stress response, such as fever and chest and back discomfort, which, in the judgment of the investigator, need not be recorded as an adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W. Zhang, Principal Investigator — Seattle，Washington，USA; Weiguo Fu, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - Jia Hu, Chengdu
  - Weiguo Fu, Shanghai
  - Honglin Dong, Taiyuan

IPD SHARING:
Plan to Share IPD: No